CLINICAL TRIAL: NCT02057653
Title: Evaluation of Goal-Directed Intraoperative Hemodynamic Optimization Protocol
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 20139795; UCIANES04 (Other: University of California, Irvine)
Record Dates: First submitted 2013-12-17; First posted 2014-02-07 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Complications
Keywords: Goal-directed fluid management
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before GDFM Training: Approximate 300 patients' medical record information will be extracted from the UC Irvine Medical Center electronic medical record prior to the start of the training curriculum.
- After GDFM Training: Approximate 300 patients' medical record information will be extracted from the UC Irvine Medical Center electronic medical record after the training program took place

SUMMARY:
As part of a quality assurance program, the Department of Anesthesiology implemented a Goal-Directed Fluid Management training course for all physicians and nurses to provide goal-directed fluid management. We intend to assess whether there has been any improvement in patient outcomes by analyzing de-identified clinical information that are readily available via the medical center electronic medical record system. The time-frame we are interested in is one year before and one year after the Goal-Directed Fluid Management training curriculum (June 15, 2011 to September 15, 2013).

DETAILED DESCRIPTION:
A number of published studies in anesthesia have demonstrated that certain patient factors may impact patient perioperative outcomes. Factors such as age, gender, cardiac function, and hemodynamic status all have been shown to be predictive indicators. The goal of the present study is to evaluate these factors with the effectiveness of the Goal Directed Fluid Management training on patient outcomes after major surgeries and document the final perioperative outcomes.

This is an observational study in which patients' de-identified clinical information will be extracted from the University of California, Irvine Medical Center electronic medical record system to evaluate whether there has been a change in patients' outcomes after the Goal-Directed Fluid Management training curriculum was implemented. We will extract data from both before and after the training took place-- the time-frame is from June 15, 2011 to September 15, 2013. Specifically we will be looking at 30 day re-admission and 90 day mortality following surgery. There are no study procedures or use of biological material. Patient identifies are utilized in the secure database as this is utilized for clinical management. When the data is extracted from the database for research purposes the patient identifiers will be removed and no patient identifiers will be included in the information during statistical analysis or subsequent reporting. For publication, only aggregate data is utilized. No identifiable patient information will be released at any time.

Statistical considerations may include: Sample Size Considerations, Predictors, Covariates/Cofounders, Statistical Goal(s), Statistical Approach, and Secondary Analysis. Specifically, statistical analysis will be performed using computerized software (SPSS for Windows version 12.0). For data that was non-normally distributed a Mann Mann-Whitney test will be used and normally distributed data will be compared using the Student T-test. Ordinal and nominal data will compared using Chi-Square analysis. A p value smaller or equal to 0.05 will be considered significant. These statistical considerations will aid in supporting the study's hypothesis for patient outcomes improvement with Early Goal Directed Fluid Management training.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older,
* Patients undergoing one or more of the following high risk surgeries: liver resection, pancreatectomy, cancer debulking, colorectal surgery,
* Surgical procedures must be projected to last longer than 2 hours,
* Patients receiving

Exclusion Criteria:

* Pregnant
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The characteristics for inclusion of the proposed subject population will include those adults patients who have undergone one or more of the following high risk surgeries: liver resection, pancreatectomy, cancer debulking, colorectal surgery, and receive arterial line as directed by the attending anesthesiologist as standard care of patient. Emergent surgical procedures will not be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The difference in length of stay in the hospital after surgery between pre-curriculum and post-curriculum cohorts. | records will be assessed an expected average of 1 year before curriculum (June 2011) and 1 year after curriculum (September 2013) June 15, 2011- September 15, 2013
  Length of stay in the hospital (number of nights) after the surgery

SECONDARY OUTCOMES:
Incidence of surgical site infection | 30 days after surgery
  Surgical site infection defined according to the NSQIP database
Incidence of postoperative pneumonia | 30 days after surgery
  Pneumonia defined according to the NSQIP database
Incidence of urinary tract infection | 30 days after surgery
  Urinary tract infection defined according to the NSQIP database
Incidence of myocardial infarction | 30 days after surgery
  Myocardial infarction defined according to the NSQIP database
Incidence of deep vein thrombosis | 30 days after surgery
  Deep vein thrombosis defined according to the NSQIP database
Incidence of atrial fibrillation | 30 days after surgery
  Atrial fibrillation defined according to the NSQIP database
Incidence of sepsis | 30 days after surgery
  Sepsis defined according to the NSQIP database
30 days readmission rate | 30 days after discharge from hospital
  Unplanned readmission within 30 days after hospital discharge.
Incidence of intraoperative transfusion | intraoperatively (Day 1, during surgery)
  Blood product transfusion during surgery
Incidence of post anesthesia care unit transfusion | 30 days after surgery in the PACU
  Blood product transfusion in the post anesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Cannesson, MD, PhD, Principal Investigator — UC Irvine Medical Center, Dept. of Anesthesiology & Perioperative Care
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Derived] Cannesson M, Ramsingh D, Rinehart J, Demirjian A, Vu T, Vakharia S, Imagawa D, Yu Z, Greenfield S, Kain Z. Perioperative goal-directed therapy and postoperative outcomes in patients undergoing high-risk abdominal surgery: a historical-prospective, comparative effectiveness study. Crit Care. 2015 Jun 19;19(1):261. doi: 10.1186/s13054-015-0945-2. PMID 26088649